CLINICAL TRIAL: NCT01603745
Title: Effects of Drospirenone-ethinylestradiol and/or NOMAC-valerate Estradiol on Cardiovascular Risk in Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zoely1984
Record Dates: First submitted 2012-05-19; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- NOMAC-valerate estradiol (Active Comparator): E/P therapy
  Interventions: Drug: Zoely
- Drospirenone/ethinylestradiol (Active Comparator): E/P therapy
  Interventions: Drug: Yasmin

INTERVENTIONS:
Drug: Zoely — 1 pill every day
  Arms: NOMAC-valerate estradiol
Drug: Yasmin — 1 pill every day
  Arms: Drospirenone/ethinylestradiol

SUMMARY:
Polycystic ovary syndrome (PCOS) is often associated with pathological conditions, such as insulin resistance (IR), type 2 diabetes (DM2), obesity and it has potentially increased risk for cardiovascular disease (CVD). Of note, risk factors for CVD including dyslipidaemia, hypertension, oxidative stress and inflammation are associated with PCOS. The investigators want to evaluate the effects of two different types of E/P therapy on cardiovascular risk in PCOS.

DETAILED DESCRIPTION:
PCOS is the most common female endocrinopathy in reproductive age. This syndrome is a heterogeneous condition characterized by several symptoms and clinical signs related to reproductive, cardiometabolic and psychological disorders.We recently demonstrated that young PCOS women show an expansion of an unusual T-cell population with proinflammatory functions, identified by CD4+CD28null T lymphocytes . Of note, this T subpopulation has been found to be expanded in patients with unstable angina, type 2 diabetes (DM2), in absence of clinical evidence of CVD 12, and has been recently associated to recurrent coronary instability .Based on the above mentioned evidences, the aim of the present study is to evaluate the effects of DRPS/EE alone versus metformin alone versus DRPS/EE plus metformin on the CD4+CD28null T cells frequency and on endocrino-metabolic parameters, in hyperinsulinemic PCOS patientsTo evaluate long-term effects of drospirenone (DRSP)/ethinylestradiol (EE) and NOMAC-valerate estardiol on some cardiovascular risk factors in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with PCOS aged 18-35 years

Exclusion Criteria:

* chronic or acute inflammatory disease
* cancer
* autoimmune disease
* treatment with clomiphene citrate
* antiandrogens
* drugs to control appetite or insulin-sensitizing drugs (metformin, pioglitazone and rosiglitazone) during the last 6 months prior to our evaluation, DM2, hypertension, major surgery in the last 3 months or other hormonal dysfunctions (hypothalamic, pituitary, thyroidal, or adrenal causes)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
cardiovascular risk | 120 minutes
  total testosterone (T), SHBG, androstenedione (A), 17-hydroxyprogesterone (17-OHP), dehydroepiandrosterone sulphate (DHEAS), triglycerides, total cholesterol, high- and low-density lipoprotein cholesterol (HDL and LDL cholesterol) and alanine aminotransferase (ALT),CD4+CD28null frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of Sacred Heart, Rome, Rome, Italy

REFERENCES:
- [Result] Niccoli G, Apa R, Lanzone A, Liuzzo G, Spaziani C, Sagnella F, Cosentino N, Moro F, Martinez D, Morciano A, Baca M, Pazzano V, Gangale MF, Tropea A, Crea F. CD4+CD28 null T lymphocytes are expanded in young women with polycystic ovary syndrome. Fertil Steril. 2011 Jun 30;95(8):2651-4. doi: 10.1016/j.fertnstert.2011.01.129. Epub 2011 Feb 16. PMID 21324454